Abbreviated Injury Scale (AIS) Grading and Simple Triage and Rapid Treatment (START) Combined with Film Transferring on Instant Message Improve The Difference of Disaster Triage and Disaster Management

NCT number: nil

date of the document: 20220414

The re-defined AIS and START grading status and primary grading documented in the medical record are compared and the Statistical methods were Spearman Rank Correlations and Wilcoxon signed rank test. The p value of statistical significance was 0.05. The regression analysis is also used to find the correlation of two groups.